CLINICAL TRIAL: NCT05279664
Title: RIC-NEC Phase II Feasibility Randomized Controlled Trial: Remote Ischemic Conditioning in Necrotizing Enterocolitis
Brief Title: RIC-NEC Randomized Controlled Trial
Acronym: RIC-NEC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Thrasher Research Fund (Other); Mount Sinai Hospital, Canada (Other); Sunnybrook Health Sciences Centre (Other); McMaster Children's Hospital (Other); Children's Hospital Medical Center, Cincinnati (Other); Children's Hospital of Orange County (Other); Karolinska University Hospital (Other); Sophia Kindergeneeskunde (Other); UCL Great Ormond Street Institute of Child Health (Other); Hospital Universitario La Paz (Other); University of Southampton (Other); Xiamen Children's Hospital, Fujian of China (Other); Shanghai Children's Hospital (Other)
Responsible Party: Principal Investigator, Agostino Pierro, Principal Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTO 3802
Record Dates: First submitted 2022-01-11; First posted 2022-03-15 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Necrotizing Enterocolitis
Keywords: remote ischemic conditioning; prematurity
MeSH Terms: conditions — Enterocolitis, Necrotizing; Premature Birth | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The intervention used in this study is remote ischemic conditioning (RIC). Patients randomized to the intervention arm will receive RIC as well as the standard medical management for NEC. RIC will consist of 4 cycles of limb ischemia (5 minutes) followed by reperfusion (5 minutes), repeated on two consecutive days. An appropriately sized blood pressure cuff (covering 2/3 of the distance between the shoulder and the elbow) will be applied by a trained research fellow or nurse to an arm (or leg if the arm is not available because of medical reasons such as central line insertion). The systolic blood pressure will be measured before the first RIC cycle using a different cuff of the same size connected to a monitor. During ischemia time, the cuff will be inflated to a pressure of 15 mmHg above the child's systolic pressure.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: RIC will be masked from the local team of healthcare workers and parents/caregivers. A trained research fellow/nurse not involved in the circle of care will perform, behind a portable sliding medical privacy screen, inflation/deflation of the cuff (RIC intervention) or sham inflation/deflation of the cuff connected to a dummy neonatal arm to mimic the noise of cuff inflation (control). Both limbs (receiving and not receiving RIC) will be blinded from the circle of care and parents/caregivers. During the RIC procedure, the research fellow/nurse will monitor the oxygen saturation of the limb receiving RIC via pulse oximetry. The circle of care will continue to monitor the neonate's clinical parameters on the cardiopulmonary monitor on the other side of the privacy screen.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (RIC + standard of care for NEC) (Experimental): Neonates randomized to the intervention arm will receive RIC and will continue to receive the standard of care for NEC.
  Interventions: Other: Remote ischemic conditioning (RIC) + Standard of Care for NEC
- Control (Standard of care for NEC) (Sham Comparator): Neonates randomized to the control arm will receive the standard of care for NEC. The research fellow or nurse responsible for performing RIC will be performing sham inflation/deflation of the blood pressure cuff connected to a dummy arm to mimic the noise of the cuff for neonates in the control arm.
  Interventions: Other: Standard of Care for NEC

INTERVENTIONS:
Other: Remote ischemic conditioning (RIC) + Standard of Care for NEC — RIC will consist of 4 cycles of limb ischemia (5 min) followed by reperfusion (5 min), repeated on two consecutive days. An appropriately sized blood pressure cuff (covering 2/3 of the distance between the shoulder and the elbow) will be applied by a trained research fellow or nurse to an arm (or leg if the arm is not available because of medical reasons such as central line insertion). The systolic blood pressure will be measured before the first RIC cycle using a different cuff of same size connected to a monitor. During ischemia time, the cuff will be inflated to a pressure of 15 mmHg above the child's systolic pressure. Neonates in this arm will continue to receive standard of care for NEC.
  Arms: Intervention (RIC + standard of care for NEC)
Other: Standard of Care for NEC — Neonates in this arm (i.e. the control arm) will receive standard of care for NEC.
  Arms: Control (Standard of care for NEC)

SUMMARY:
Necrotizing enterocolitis (NEC) is a serious intestinal disease of preterm and term neonates which remains a major cause of intestinal failure, and an unsolved clinical challenge in pediatrics. While overall mortality of preterm infants continues to decrease due to improvements in general neonatal care, mortality caused by NEC remains high (up to 30-50%) and survivors suffer from reduced quality of life, and long-term disabilities such as debilitating complications of intestinal failure, poor growth and neurodevelopmental delay. Besides prevention, there have been hardly any innovations in the treatment of NEC which underwent trial evaluation.

NEC pathogenesis is multifactorial, but bowel ischemia is known to play an essential role in the development of NEC. Remote ischemic conditioning (RIC) is a therapeutic maneuver that involves brief cycles of non-lethal ischemia and reperfusion applied to a limb, which protects distant organs (such as the intestine) from ischemic damage. The investigators have shown that in preclinical models of NEC, RIC effectively reduces intestinal damage and prolongs survival. The investigators have also demonstrated the safety of RIC in preterm neonates with NEC. Before the investigators can evaluate the effectiveness of RIC in treating neonates with NEC in a Phase III randomized clinical trial (RCT), a Phase II Feasibility RCT must be conducted to evaluate issues related to the enrollment and randomization of neonates, masking of the RIC intervention, and measurement of clinical outcomes.

The investigators hypothesize that it is feasible to conduct a multicenter RCT to evaluate RIC during the management of neonates with medical NEC.

DETAILED DESCRIPTION:
Background: Necrotizing enterocolitis (NEC) is a serious intestinal disease of preterm and term neonates which remains a major cause of intestinal failure, and an unsolved clinical challenge in pediatrics resulting in mortality rates as high as 50%, reduced quality of life and long-term disabilities such as short bowel syndrome, poor growth, and neurodevelopmental delay. Experimentally, the investigators have discovered that intestinal and brain damage, as well as mortality following NEC, can be avoided by remote ischemic conditioning (RIC) in the early stage of the disease. Remote ischemic conditioning is a therapeutic maneuver involving brief cycles of non-lethal ischemia and reperfusion applied to a limb that protects distant organs (such as the intestine) from sustained ischemic damage. In the clinical setting, the cycles of ischemia and reperfusion can be administered by inflation and deflation of a blood pressure cuff, similar to routine blood pressure measurements. The investigators have also demonstrated that this non-invasive, simple, and easy-to-use maneuver consisting of inflation/deflation of a blood pressure cuff on the upper arm is safe in preterm human neonates with NEC.

Hypothesis and Objectives: The investigators hypothesize that a masked multi-center randomized controlled trial of RIC in neonates with early-stage NEC is feasible.

Study design: This is a Phase II multicenter, masked, randomized controlled feasibility trial consisting of two arms: RIC (intervention) and no RIC (control).

Study population: Preterm neonates with clinical and radiological evidence of early-stage NEC and receiving medical treatment.

Sample size/power of primary endpoint: In the 12 international collaborating centers, the investigators expect to randomize, in 30 months, 78 patients with NEC receiving medical treatment (39 per arm) which represents 40% of approached eligible neonates.

ELIGIBILITY:
Inclusion Criteria:

1. All gestational age at birth.
2. Current weight ≥600 g
3. Confirmed diagnosis of "medical" NEC based on the joint opinion of two attending experts in the field (two neonatologists or one neonatologist and one pediatric surgeon).
4. NEC diagnosis established within the previous 24 hours.

Exclusion Criteria:

1. Indication for surgery in the joint opinion of the attending neonatologist and pediatric surgeon (i.e. surgical NEC). This diagnosis is based on the presence of pneumoperitoneum in the abdominal radiograph and/or failure of medical treatment for NEC
2. Previous episodes of NEC
3. Diagnosis of NEC established >24 hours ago
4. Major congenital heart disease which needs surgical repair
5. Antecedent limb ischemia/limb thrombotic events, occlusive arterial or venous thrombosis
6. Associated gastrointestinal anomalies including gastroschisis or congenital diaphragmatic hernia.

Min Age: 0 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2025-12-20 (Actual); Study Completion 2026-03-18 (Estimated)

PRIMARY OUTCOMES:
The proportion (% total) of screened patients that are eligible for enrollment in the trial. | 24 hours
  The investigators will determine the proportion (% total) of screened patients who meet the inclusion criteria and do not meet the exclusion criteria and are therefore eligible for enrollment in this study.
The proportion (% total) of eligible patients that give consent and are randomized. | 24 hours
  The investigators will determine the proportion (% total) of eligible patients for whom informed consent from parents/caregivers can be obtained and randomization can be completed within 24 hours from confirmed diagnosis of medical NEC by a neonatologist and pediatric surgeon.
The proportion (% total) of randomized patients that receive allocated intervention. | 72 hours
  The investigators will determine the proportion (% total) of patients randomized to each study arm who successfully receive the intervention corresponding to that arm: RIC or no RIC.
The proportion (% total) of randomized patients receiving masked allocated intervention. | 72 hours
  The investigators will determine the proportion (% total) of randomized patients that receive the allocated intervention (RIC or no RIC) successfully masked from the circle of care as well as parents/caregivers.
The proportion (% total) of randomized patients assessed for NEC-related outcomes. | 3 months +/- 1 week
  The investigators will determine the proportion (% total) of randomized patients that are successfully assessed for the NEC-related outcomes (please see secondary outcomes 6-13 below).

SECONDARY OUTCOMES:
Number of patients surviving without the development of intestinal perforation, necrosis or stricture. | 3 months +/- 1 week
  The investigators will determine the number of randomized patients who survive at 1 month and 3 months post-randomization without developing intestinal perforation, intestinal necrosis, or intestinal stricture.
Timing and cause of death | 3 months +/- 1 week
  The time, and if possible, the cause of death will be recorded during the 90 days post-randomization considering whether it was possible to determine if death was related to complications of NEC or to a disease process in other systems including cardiac, neurological, respiratory, renal, metabolic.
Number, type and times of abdominal operations performed. | 3 months +/- 1 week
  The number, time(s), and type(s) of abdominal operations (insertion of peritoneal drainage or laparotomy) performed during the 90 days post-randomization will be recorded.
Number of patients receiving parenteral nutrition | 3 months +/- 1 week
  The number of patients receiving parenteral nutrition during the 90 days post-randomization will be recorded as a measure of intestinal function.
Number of patients developing severe neurological injury | 3 months +/- 1 week
  Development of severe neurological injury will be assessed based on head ultrasound at 1-month and 3-months post-randomization and will be defined as the presence of intraventricular hemorrhage (IVH), ventricular enlargement, parenchymal echogenicity or periventricular leucomalacia (PVL).
Number of patients developing chronic lung disease (CLD) | 3 months +/- 1 week
  Development of chronic lung disease (CLD) during the 90 days post-randomization will be defined as respiratory support given at 36 weeks' postmenstrual age or at discharge (if earlier than 36 weeks' postmenstrual age) to level 2 neonatal intensive care unit (NICU) and classified in different degrees of severity from mild to moderate to severe CLD according to the criteria published in the Canadian Neonatal Network (CNN) Annual Report (2019).
Number of patients developing severe retinopathy of prematurity (ROP) | 3 months +/- 1 week
  During the 90 days post-randomization, the investigators will assess the development of Stage 3, 4 or 5 retinopathy of prematurity (ROP) as defined by the International Classification of ROP and/or those infants requiring treatment (laser or intraocular injection). ROP will be scored as the highest stage in either eye identified at any time.
Survey of stakeholders' satisfaction | 1 month +/- 1 week
  Satisfaction of key trial stakeholders (parents and healthcare workers) with the recruitment process, delivery and masking of the intervention will be evaluated by questionnaires, using a scale of 0-4. Higher scores indicate greater satisfaction and lower scores indicate less satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Agostino Pierro, OBE, MD, Principal Investigator — The Hospital for Sick Children
Locations (4):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States
- Canada (3):
  - Sunnybrook Health Sciences Center, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koike Y, Li B, Ganji N, Zhu H, Miyake H, Chen Y, Lee C, Janssen Lok M, Zozaya C, Lau E, Lee D, Chusilp S, Zhang Z, Yamoto M, Wu RY, Inoue M, Uchida K, Kusunoki M, Delgado-Olguin P, Mertens L, Daneman A, Eaton S, Sherman PM, Pierro A. Remote ischemic conditioning counteracts the intestinal damage of necrotizing enterocolitis by improving intestinal microcirculation. Nat Commun. 2020 Oct 2;11(1):4950. doi: 10.1038/s41467-020-18750-9. PMID 33009377
- [Background] Chen Y, Koike Y, Chi L, Ahmed A, Miyake H, Li B, Lee C, Delgado-Olguin P, Pierro A. Formula feeding and immature gut microcirculation promote intestinal hypoxia, leading to necrotizing enterocolitis. Dis Model Mech. 2019 Dec 9;12(12):dmm040998. doi: 10.1242/dmm.040998. PMID 31704804
- [Background] Chen Y, Chang KT, Lian DW, Lu H, Roy S, Laksmi NK, Low Y, Krishnaswamy G, Pierro A, Ong CC. The role of ischemia in necrotizing enterocolitis. J Pediatr Surg. 2016 Aug;51(8):1255-61. doi: 10.1016/j.jpedsurg.2015.12.015. Epub 2016 Jan 8. PMID 26850908
- [Background] Alganabi M, Lee C, Bindi E, Li B, Pierro A. Recent advances in understanding necrotizing enterocolitis. F1000Res. 2019 Jan 25;8:F1000 Faculty Rev-107. doi: 10.12688/f1000research.17228.1. eCollection 2019. PMID 30740215
- [Background] Neu J, Walker WA. Necrotizing enterocolitis. N Engl J Med. 2011 Jan 20;364(3):255-64. doi: 10.1056/NEJMra1005408. No abstract available. PMID 21247316
- [Background] Willan AR, Thabane L. Bayesian methods for pilot studies. Clin Trials. 2020 Aug;17(4):414-419. doi: 10.1177/1740774520914306. Epub 2020 Apr 16. PMID 32297539